CLINICAL TRIAL: NCT05448339
Title: The Value of Tumor Feeding Vessels Deprivation Combined With Tyrosine Kinase Inhibitor in Liver Transplantation
Brief Title: Tumor Feeding Vessels Deprivation Combined With Tyrosine Kinase Inhibitor in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Lin Zhong, director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHLTQC-5
Record Dates: First submitted 2022-06-29; First posted 2022-07-07 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVHA: Patients undergo tumor feeding vessels deprivation
  Interventions: Combination Product: PVHA or TACE
- TACE: Patients undergo TACE therapy
  Interventions: Combination Product: PVHA or TACE

INTERVENTIONS:
Combination Product: PVHA or TACE — PVHA or TACE

SUMMARY:
To investigate the value of tumor feeding vessels deprivation combined with tyrosine kinase inhibitor in liver transplantation. Patients are enrolled into two groups according to the downstaging therapy they undergo before transplantion.

ELIGIBILITY:
(1) age ≥18 years; (2) exceeding UCSF criteria; (3) absence of vascular invasion, nodal involvement, or extrahepatic metastases; (4) receiving TACE treatment or LTFVD treatment for downstaging purposes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) age ≥18 years; (2) exceeding UCSF criteria; (3) absence of vascular invasion, nodal involvement, or extrahepatic metastases; (4) receiving TACE treatment or LTFVD treatment for downstaging purposes. Patients who underwent resection, LT, or any form of downstaging treatment prior to enrollment were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Underwent LT | January 2013 and December 2020
  Underwent LT
Successful downstaging | January 2013 and December 2020
  Successful downstaging

SECONDARY OUTCOMES:
AFP reduction of patients | January 2013 and December 2020
  AFP reduction of patients
Survival time of patients | January 2013 and December 2020
  Survival time of patients
Recurrence of patients | January 2013 and December 2020
  Recurrence of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No